CLINICAL TRIAL: NCT02022475
Title: Effect of Peroral Vitamin D Versus Placebo on Self-reported Fatigue in Adults With Low 25-hydroxy-vitamin D Levels
Brief Title: Effect of Vitamin D Treatment on Fatigue
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kray-1213
Record Dates: First submitted 2013-12-12; First posted 2013-12-27 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; fatigue
MeSH Terms: conditions — Vitamin D Deficiency; Fatigue | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Active Comparator): 100 000 units vitamin D3 single dose
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): similar appearance
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Vitamin D — 100 000 units oral vitamin D as 2 capsules 50 000 units each
  Other Names: Cholecalciferol
  Arms: Cholecalciferol
Other: placebo — 2 placebo capsules will be applied as a single dose
  Arms: Placebo

SUMMARY:
Primary objective

-Change in Fatigue Assesment Score (FAS) between the first visit (baseline) and 28 (+maximum 7) days after oral administration of 100 000 E vitamin D (Cholecalciferol).

Secondary objectives

* Effect of oral administration of vitamin D on serum vitamin D levels (25-Hydroxy-Vitamin D = Colecalciferol), PTH, Calcium, and Phosphate as compared to placebo.
* Efficacy of vitamin D (Colecalciferol) administration on fatigue using the short self-developed FCA-Test
* Safety of 100 000 E oral vitamin D (Colecalciferol) administration as compared to oral placebo. Laboratoty parameters such as serum calzium and phosphate levels and the number of adverse events compared to placebo will be used for safety monitoring.
* Efficacy of oral administration of vitamin D (Cholecalciferol) on plasma FGF-23, Sclerostin and Klotho levels compared to placebo.

DETAILED DESCRIPTION:
1. General Design

   This is a randomized, double blind, mono-centric, placebo-controlled interventional study of the effects of oral vitamin D supplementation on self-reported fatigue. Overall 80 patients with proven vitamin D deficiency (20-Hydroxy-Vitamin D ≤ 20 µg/L) who fulfill all the eligibility criteria will be randomized and enrolled to receive vitamin D or placebo in 1:1 ratio. All patients must sign an informed consent prior to enrolment and meet eligibility criteria. All patients will be recruited at the Medical Outpatients Department of University Hospital Zürich.

   Screening, Part 1: Consecutive patients consulting the Medical Outpatients Department, complaining of fatigue, will be asked to participate in the study. Basic questionnaire for fatigue will be applied to confirm fatigue symptoms.

   Screening, Part 2: In positive case, the patients will be asked to sign an informed consent. Beck Depression Inventory (BDI), Mini International Neuropsychiatric Interview (M.I.N.I.) and Insomnia Severity Index (ISI) will be administered to exclude depression, sleep disorders and major psychiatric disorders respectively. Thereafter blood will be tested according to table 1. Patients with vitamin D levels below 20 µg/L will undergo randomization. Participants will be informed about their results of vitamin D levels by the telephone, a treatment appointment within 2 weeks after screening will be arranged for participants with vitamin D levels ≤ 20 µg/L.

   Visit A (within 2 weeks after randomisation): Routine clinical examination will be performed. Baseline Fatigue assessment scale (FAS) score will be documented, following by blood and urine samples according to table 1 to measure the baseline vitamin D-, PTH- and Calcium levels. Blood samples will undergo centrifugation. Blood and urine samples will be frozen at -80°C.

   Oral Vitamin D preparation or placebo will be administered according to the protocol in a double blinded manner. The drug administration will be done by an independent person e.g. a physician assistant or study nurse directly observing the drug intake. During the administration, procedures are implemented which ensure that the subjects cannot distinguish between placebo and verum (identical appearance, taste and smell).

   Visit B ( 4 weeks after Visit A + maximum 7 days): Patients will undergo the same Assessment of Fatigue by filling out FAS questionnaire. Additionally, a short self-developed test Fatigue course assessment (FCA) will be applied to evaluate symptomatic response. Thereafter blood and urine samples will be taken to document biochemical response: Vitamin D-, PTH-, phosphate and calcium levels.

   The Vitamin D status of the subjects will be monitored by standard clinical chemical parameters. Safety assessments will include pre- and post-treatment measurement of vital signs, clinical laboratory assessments, and the recording of adverse clinical events.
2. Selection of study population / Subject recruitment

   Patients will be informed about the study at a regular medical visit at the medical outpatients department USZ. Potential subjects will be provided with the participant information sheet and fill in the basic questionnaire for fatigue.

   After informed consent has been obtained, all study-specific information will be collected to determine if a patient meets the inclusion criteria without violating any of the exclusion criteria. A total number of 80 subjects will be enrolled, with an enrolment goal of 12 subjects per month. Recruitment will take place in the medical outpatient department (Klinik und Poliklinik für Innere Medizin) of the University Hospital in Zurich. If monthly enrolment goals cannot be achieved, announcements will be posted on the university's announcement boards and on the internet page of the USZ medical department. Patients will receive no financial compensation.

   The specific inclusion and exclusion criteria for enrolling subjects in this study are described in the following sections.
3. Prior and Concomitant Therapy

   According to the inclusion/exclusion criteria (see above), chronic intake of concomitant medication is not allowed, except oral contraceptives. Intake of Vitamin D preparations during the last 8 weeks before the start of the trial protocol and during the trial is not allowed. Vitamin preparations or herbal medicine should be withheld during the study period.

   Sporadic medication with e.g. NSAID or paracetamol for symptomatic treatment of intercurrent viral infections or occasional headaches is allowed. All concomitant medications have to be recorded on the CRF. Subjects taking additional vitamin D preparations drugs the study course will be excluded from the study.
4. Randomization and blinding

   Overview:

   A randomization procedure will be used to avoid a bias in the assignment of the study subjects to the two treatment groups (oral vitamin D, oral placebo). Randomization lists, preparation of study drugs and placebo, labelling and drug accountability will be done by the hospital pharmacy (Kantonsapotheke Zürich). The randomisation list will be preserved by the hospital pharmacy. The oral intake will be directly observed by a physician assistant or study nurse. As placebo and verum are manufactured having identical appearance, taste and smell, study participants can not differ between placebo and verum.

   Procedure:

   Patients will be assigned to treatment groups based on a randomization list/schedule prepared by the hospital pharmacy prior to the trial. Patients will receive a randomization number. Randomized patients who terminate their study participation for any reason regardless whether the study medication was taken or not, will retain their randomization number. The next patient will be given the next randomization number.

   An Emergency Code Break preserved in a sealed Emergency Code Envelope will be available to the investigator. This envelope with the Code Break should only be opened in emergency situations when the identity of the investigational product must be known by the investigator in order to provide appropriate medical treatment.
5. Treatment / Dosage and administration

The patients will be randomized to one of the 2 treatment groups (40 participants in each group): Group I: oral vitamin D; Group II: oral placebo.

* Group I (oral vitamin D): 100 000 E Vitamin D (Colecalciferol) will be applied as a single dose as two capsules containing 50 000 E each.
* Group II (oral placebo): 2 placebo capsules will be applied as a single dose The drug preparations will be delivered and labelled by the hospital pharmacy according to standard operating procedures and GMP guidelines.

After the study finalisation, the placebo group will be offered a treatment with Vitamin D.

5. Study drug information Vitamin D used in this study is 2 capsules containing 50 000 E Cholecalciferol each, prepared by the university hospital pharmacy.

Placebo will be prepared by the university hospital pharmacy in a capsule of identical appearance, taste and smell.

6. Packing and Labeling Study medication (oral Vitamin D and placebo) will be provided by the hospital pharmacy, labelled and packaged according to Swiss guidelines and EU-GMP guidelines.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-25 kg/m2
* Serum 25-Hydroxy-Vitamin D level < 20 mkg/l
* Adequate contraception during the study period
* Informed consent

Exclusion Criteria:

* Anemia with Hb level < 120 g/l
* Known hypersensitivity to vitamin D
* Intake of vitamin D preparations (including) during the last 8 weeks before the start of the trial protocol
* Pregnancy or lactation or intention to become pregnant during the course of the study
* Any cardiovascular, pulmonary, renal or hepatic disease
* Presence of muscle disease, CK>167 U/L
* Presence of known bone disease, alkaline phosphatase > 104 U/l
* Severe infection/inflammation or malignancy
* Known mental disorders (e.g. depression), sleep disorders
* Chronic intake of concurrent medication, except oral contraceptives. Sporadic intake of NSAID or paracetamol, e.g. in the case of a common cold or sporadic headaches is allowed.
* CRP > 10 mg/l
* TSH out of normal range
* Ferritin <15 µg/L
* Any concurrent medical condition(s) that, in the view of the investigator, would prevent compliance or participation or jeopardize the health of the participants.
* Participation in any other therapeutic trial within the previous month
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia etc.
* Enrollment of the investigator, his/her family members, employees and other dependent persons

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Intraindividual change of Fatigue as quantified by FAS (δFAS) 28 (+maximum 7) days after administering Vitamin D3 (Cholecalciferol) | 28 (+maximum 7) days

SECONDARY OUTCOMES:
Efficacy of oral administration of vitamin D on serum vitamin D levels (25-Hydroxy-Vitamin D = Cholecalciferol), PTH, Calcium, and Phosphate as compared to placebo. | 28 (+maximum 7) days
  Blood samples will be drawn, urine samples will be taken prior to and 28 (+maximum 7) days after the vitamin D administration.

OTHER OUTCOMES:
Efficacy of vitamin D (Cholecalciferol) administration on fatigue using the short self-developed FCA-Test | 28 (+maximum 7) days
  Fatigue course assessment (FCA)
  Wie würden Sie ihre momentane Müdigkeit/Erschöpfung im Vergleich zur Situation vor der Behandlung beschreiben?
  Beschwerdefrei Besser Unverändert Schlechter Deutlich schlechter
Fibroblast Growth factor 23, sclerostin and soluble Klotho levels before and 28 days after vitamin D administration | 28 (+maximum 7) days

CONTACTS AND LOCATIONS:
Overall Officials: Krayenbühl Pierre-Alexander, Dr, Study Director — University Hospital Zürich, Department of Internal Medicine; Albina Nowak, MD, Principal Investigator — University Hospital Zürich, Department of Internal Medicine
Locations (1):
- Clinic and policlinic for Inetrnal Medicine, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Nowak A, Boesch L, Andres E, Battegay E, Hornemann T, Schmid C, Bischoff-Ferrari HA, Suter PM, Krayenbuehl PA. Effect of vitamin D3 on self-perceived fatigue: A double-blind randomized placebo-controlled trial. Medicine (Baltimore). 2016 Dec;95(52):e5353. doi: 10.1097/MD.0000000000005353. PMID 28033244